CLINICAL TRIAL: NCT00816322
Title: The Effect of Fish Oil in Major Depressive Disorder: a Double-blind Placebo-controlled Monotherapy Trail and a RCT for Recurrence Prevention
Brief Title: The Effect of Fish Oil in Major Depressive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, Kuan-Pin, Researcher, National Science and Technology Council, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DMR93-IRB-87
Record Dates: First submitted 2008-12-31; First posted 2009-01-01 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- omega-3 fatty acids (Active Comparator): EPA 2.1 g/d+DHA 1.1 g/d
  Interventions: Dietary Supplement: Omega-3 fatty acids
- Placebo (Placebo Comparator): high oleic oil
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Omega-3 fatty acids — EPA 2.1 g/d+DHA 1.1 g/d
  Arms: omega-3 fatty acids
Dietary Supplement: Placebo — high oleic oil
  Arms: Placebo

SUMMARY:
The whole study was divided into two major parts: (A) the 12-week, double-blind, randomized controlled, parallel omega-3 fatty acid monotherapy study in 60 patients with mild to moderate major depressive disorder. (B) The double-blind, randomized controlled, parallel omega-3 fatty acid add-on prevention study in 60 patients with major depressive disorder in recovery status.

The goals of this study were to examine the therapeutic and recurrence prevention effects of omega-3 fatty acids on major depressive disorder.

ELIGIBILITY:
Inclusion Criteria:

1. DSM-IV criteria for major depressive disorder.
2. Age being age 18-65.
3. Capacity and willingness to give written informed consent.

Exclusion Criteria:

1. Any major medical illnesses.
2. A recent or past history of any Axis-I diagnoses besides major depressive disorder, including psychotic disorders; cognitively impaired mental disorders; impulse control disorders; substance use disorder or substance abuse (last 6 months prior to the studies); primary anxiety disorders, including post-traumatic stress disorder and panic disorder; and bipolar disorders; or Axis-II diagnoses, i.e. borderline and antisocial personality disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2005-01; Primary Completion 2014-01 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
HAMD | W0 W2 W4 W8 W12

SECONDARY OUTCOMES:
BDI | W0 W2 W4 W8 W12
Adverse effects | W0 W2 W4 W8 W12
Recurrence rate | M0 M1 M2 M3 M4 M6

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University, Taichung, Taichung, Taiwan

REFERENCES:
- [Derived] Appleton KM, Voyias PD, Sallis HM, Dawson S, Ness AR, Churchill R, Perry R. Omega-3 fatty acids for depression in adults. Cochrane Database Syst Rev. 2021 Nov 24;11(11):CD004692. doi: 10.1002/14651858.CD004692.pub5. PMID 34817851